CLINICAL TRIAL: NCT00146042
Title: Phase II Study of Tailored-Dose Docetaxel + Trastuzumab in Her-2 Positive Metastatic Breast Cancer
Brief Title: UMCC 9901: Phase II Study of Tailored-Dose Docetaxel + Trastuzumab in Her-2 Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9901; H1880n
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: HER-2 Positive Metastatic Breast Cancer
MeSH Terms: interventions — Docetaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel
Drug: Trastuzumab
Procedure: Erythromycin Breath Test (ERMBT)

SUMMARY:
This is a research study which aims to improve the way that doctors determine the dose of chemotherapy given to patients. Right now, chemotherapy is determined by a patient's height and weight. However, some patients metabolize chemotherapy faster or slower than the average person because of a different level of drug metabolizing enzyme in the liver. Therefore, some patients are either given too small or too large a dose of chemotherapy because the amount of enzyme is not taken into account. This research study will examine the use of a simple test, call the Erythromycin Breath Test(ERMBT) to determine the amount of enzyme which can metabolize the chemotherapy drug docetaxel (Taxotere). The dose of docetaxel will be tailored to the amount of enzyme which is available to metabolize the drug for each patient. The drug, docetaxel, is combined with another drug, trastuzumab (Herceptin), because at this time this combination appears to be promising in metastatic breast cancer research.

DETAILED DESCRIPTION:
This is a research study which aims to improve the way that doctors determine the dose of chemotherapy given to patients. Right now, chemotherapy is determined by a patient's height and weight. However, some patients metabolize chemotherapy faster or slower than the average person because of a different level of drug metabolizing enzyme in the liver. Therefore, some patients are either given too small or too large a dose of chemotherapy because the amount of enzyme is not taken into account. This research study will examine the use of a simple test, call the Erythromycin Breath Test(ERMBT) to determine the amount of enzyme which can metabolize the chemotherapy drug docetaxel (Taxotere). The dose of docetaxel will be tailored to the amount of enzyme which is available to metabolize the drug for each patient. The drug, docetaxel, is combined with another drug, trastuzumab (Herceptin), because at this time this combination appears to be promising in metastatic breast cancer research.-Patients participating in this study will have biopsy proven, measurable metastatic breast cancer.

During the study:

* Patients will receive tailored-dose docetaxel and Trastuzumab for their breast cancer.
* There are no sex or age restrictions although the patients in this disease category are reflective of an adult female population.

Approximately 30 subjects will be recruited at this site.

Diagnosis and Staging • All patients will have primary tumor measurements by physical exam and/or radiographic studies (CT, MRI, bone scan).

Erythromycin Breath Test*

• The ERMBT will be administered in the outpatient setting, prior to the first cycle of docetaxel. Twenty minutes after the injection of a trace amount of (14C N-methyl) erythromycin, (This test assesses the activity of the cytochrome P450 enzyme which is largely responsible for the metabolism of the chemotherapeutic agent docetaxel.)patients will exhale through a tube creating bubbles in a solution of hyamine hydroxide, ethanol, and a blue indicator until 2 mmol of carbon dioxide has been trapped and the blue color vanishes.

Chemotherapy Regimen

Premedications

* Dexamethasone 8 mg po bid for three days, beginning the day prior to docetaxel administration.
* Diphenhydramine 50 mg IVPB
* Granisetron 2 mg po 30 minutes pre-docetaxel

Chemotherapy

* Docetaxel, tailored dose, to be infused over 1 hour on day 1 every 3 weeks for the duration of study.
* Starting dose of docetaxel to be determined by the ERMBT and serum albumin according to formula as stated in protocol (page 11).
* Trastuzumab, 4 mg/kg to be infused over 90 minutes on day 2 (after pharmacokinetic sampling).
* Beginning week 2, trastuzumab will be given at a dose of 2 mg/kg weekly throughout duration of study. (After the first dose of docetaxel, future doses may be given on the same day as docetaxel).

Suggested post-chemotherapy antiemetics:

* Compazine 10 mg po q 6 hours prn nausea/vomiting Pharmacokinetic Analysis
* All patients will have pharmacokinetic determination with blood drawn for pharmacokinetic analysis over a 24 hour period after the first docetaxel treatment. Time points include time 0, 15 minutes, 45 minutes, 180 minutes (3 hours), 390 minutes (6.5 hours), and 1440 minutes (24 hours).

DEXA Scan*

* DEXA scan will be performed during the patient's stay in the Clinical Research Center, on the Lunar DPXL Bone Densitometer. This is a very simple and noninvasive test which uses x-rays and a computer program to analyze the ratio of 38 keV to 70 keV attenuation. The program then calculates Fat and Lean values for the arms, legs, abdomen, ribs, and the total body. This is the same test that is in widespread clinical use for the evaluation of osteoporosis. During the DEXA scan, patients will be exposed to a trace amount of radiation which is equal to about 2% of the yearly background dose, or less.

  *The amount of radiation to be administered by the erythromycin breath test and DEXA scan is not medically significant.
* Patients will receive 2 cycles of docetaxel/trastuzumab and be re-evaluated for response (ever 6 weeks, or later if dosage delays caused lengthening of cycle).
* Responding and stable patients will continue to receive docetaxel therapy, with evaluations every 2 cycles (every 6 weeks, or later if dosage delays caused lengthening of cycle).
* Continued treatment beyond 8 cycles will be at the discretion of the patient's primary oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven, measurable metastatic breast cancer. Patients with bone-only, and/or effusion-only disease are excluded.
* HER-2 neu positive by standard immunohistochemical criteria (2+ positivity).
* No prior chemotherapy for distant metastatic disease.
* Prior paclitaxel in the adjuvant setting is allowed.
* Karnofsky performance status equal to 70 or greater.
* ANC > 1500, Hgb > 10, plt > 100.
* Patients with some degree of hepatic dysfunction and renal dysfunction are encouraged, in order to evaluate the ability of the ERMBT in tailoring dose in these patient populations.

Exclusion Criteria:

* Age less than 18 years.
* Allergy to erythromycin.
* Previous treatment with docetaxel. Prior paclitaxel is allowed.
* Grade > 2 peripheral neuropathy.
* No confounding factors present to provide misinterpretation of data (i.e., concurrent malignancy).
* Patients who are pregnant or nursing will not be eligible for this protocol. Women of childbearing age who are not practicing reliable birth control must have a documented negative serum HCG.
* Patients who require concurrent treatment with drugs which are known to induce or inhibit CYP3A activity will be ineligible for the trial. This list includes the drugs midazolam, anti-mycotic agents (ketoconazole and related compounds), macrolide antibiotics (erythromycin and related compounds), nifedipine, anti-seizure drugs, and rifampin (induction).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1999-03; Primary Completion 2004-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To assess whether assignment of docetaxel dose based on the ERMBT will result in decreased variability in drug area under the curve when compared to dosing based on body surface area. | 2 months

SECONDARY OUTCOMES:
• To evaluate the safety and efficacy of tailored-dose docetaxel + trastuzumab in HER-2 neu positive women as first-line treatment in metastatic breast cancer. | 3 months
• To evaluate the efficacy of tailored-dose docetaxel + trastuzumab in HER-2 neu positive women, in terms of response rate and time to progression. | 6 months
• To explore the relationship between response to therapy and HER-2 status by differential polymerase chain reaction (PCR) vs. protein immunohistochemistry. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Schott, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States